CLINICAL TRIAL: NCT06994364
Title: Efficacy of Psoas Muscle Release in Young Adults With Non-specific Mechanical Low Back Pain: Randomized Controlled Trial
Brief Title: Psoas Muscle Release in Non-specific Mechanical Low Back Pain
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Escola Superior de Tecnologia da Saúde do Porto (Other)
Responsible Party: Principal Investigator, Natália Maria Oliveira Campelo, Doctor teacher, Escola Superior de Tecnologia da Saúde do Porto
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: OST1- 017
Record Dates: First submitted 2025-05-20; First posted 2025-05-29 (Actual); Last update posted 2025-09-16 (Actual); Status verified 2025-09

CONDITIONS: Low Back Pain
MeSH Terms: conditions — Low Back Pain

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Control group (Placebo Comparator): In the control group, the simulation of the technique for listening to the mobility and motility of the small intestine was performed by placing one hand on the abdomen, without pressure.
  Interventions: Other: Simulation of the intestinal listening technique.
- Experimental group (Experimental): In the experimental group, the trigger point release technique for the psoas muscle was performed.
  Interventions: Other: Trigger point release

INTERVENTIONS:
Other: Trigger point release — Ischemic compression technique is based on the application of manual pressure to treat trigger points.
  The patient was asked to lie in the supine position on the examination table. The osteopath identified the muscle through deep palpation and movement-based muscle differentiation, then applied 90 seconds of tolerable pressure to the trigger point on both sides.
  Arms: Experimental group
Other: Simulation of the intestinal listening technique. — The patient will be asked to lie in a supine position on the treatment table to simulate the listening technique for assessing the mobility and motility of the small intestine without influencing the final results, with the sensory hand placed below the umbilicus.
  Arms: Control group

SUMMARY:
Nonspecific low back pain affects approximately 80% of the population at some point in their lives.

The psoas muscle-positioned between the lumbar and pelvic regions-together with the paravertebral muscles, constitutes the primary muscular group responsible for dynamic stabilization of the spine. Alterations in this muscle may contribute to the onset of low back pain by modifying spinal biomechanics, particularly through increased lumbar lordosis and greater mechanical overload in the lumbar region.

Latent myofascial trigger points are asymptomatic but can lead to muscle shortening and weakness. They are characterized by local tenderness and may provoke a localized muscular response known as a local twitch response.

The aim of this randomized experimental study was to evaluate the immediate effect of ischemic compression applied to the trigger point of the psoas muscle on pain perception and lumbar range of motion.

Researchers will compare a group with a placebo technique to see if the release of the psoas muscle produces effects in this condition.

The variables analyzed in this study included low back pain, assessed using the Numeric Pain Rating Scale (NPRS); lateral lumbar flexion (right and left), measured using a tape measure (distance from the third finger to the floor); and lumbar flexion range of motion, assessed using the Schober test.

DETAILED DESCRIPTION:
The present study will be a randomized, double-blind clinical trial designed to analyze the immediate effect of trigger point release of the psoas muscle on pain and lumbar spine range of motion in young adults with nonspecific mechanical low back pain.

The research will involve a sample composed of individuals aged between 18 and 30 years, who will have experienced low back pain within one month prior to participation and will present a latent trigger point in the psoas muscle.

Participants will be randomly assigned to two groups: the experimental group, which will undergo the ischemic compression technique on the psoas muscle; and the control group, which will receive a simulated technique involving listening to the mobility and motility of the small intestine. Assessments will be conducted before and after the intervention using the Visual Analog Scale (VAS), the Numeric Pain Rating Scale (NPRS), measurement of lumbar lateral flexion with a measuring tape, and the modified Schober test for trunk forward flexion.

This study will aim to address the existing gap in the literature regarding the effectiveness of specific osteopathic techniques applied to the psoas muscle in relieving low back pain and improving mobility and range of motion. The methodological rigor, randomization, and double-blind design will contribute to ensuring the reliability of the collected data and the validity of the results obtained.

ELIGIBILITY:
Inclusion Criteria:

* Age between 18 and 30 years.
* Presence of low back pain for less than 1 month.
* Presence of a latent trigger point in the psoas muscle.

Exclusion Criteria:

* Volunteers with low back pain caused by: Disc herniation, Tumor, Infection, Fracture, Osteoporosis, Structural deformity or Inflammation.
* Individuals with a history of spinal surgery.
* Continuous use of analgesics.
* Participants who had undergone manual therapy in the previous month.
* Pregnant individuals.
* Obese individuals.
* Students of Osteopathy (from the 2nd, 3rd, or 4th year) and professionals in the manual therapy field.
* Participants presenting red flags for osteopathic intervention.
* Individuals with cognitive impairments that hindered their ability to understand the study/project.

Ages: 18 Years to 30 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 40 (Estimated)
Dates: Start 2026-04 (Estimated); Primary Completion 2026-08 (Estimated); Study Completion 2026-09 (Estimated)

PRIMARY OUTCOMES:
Low back pain | Immediately after the intervention
  Low back pain was evaluated using the Numeric Pain Rating Scale (NPRS), a widely used unidimensional instrument for assessing pain intensity in adults. The NPRS is a segmented numeric adaptation of the Visual Analogue Scale (VAS), consisting of a horizontal bar with 11 points, where values range from 0 ("no pain") to 10 ("worst imaginable pain").
  Each participant was asked by the researcher to indicate the number, from 0 to 10, that best represented their pain level.
Range of motion | Immediately after the intervention
  Lumbar lateral flexion was assessed using a measuring tape to evaluate the distance from the third fingertip to the floor, while lumbar flexion was measured using the Modified Schober Test.
  For lateral flexion, the participant stood upright and performed lateral flexion to the right, with the evaluator measuring the distance from the third finger to the floor. The same procedure was repeated for the left side.
  The Modified Schober Test was used to assess lumbar flexion. With the participant standing, the evaluator identified the posterior superior iliac spines (PSIS) and marked a point 15 cm above it. The participant then performed maximal forward trunk flexion with knees extended, and the distance between the two marks was measured.
  Lumbar flexion range was the difference between the initial 15 cm and the measurement after flexion.

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Furtado RN, Ribeiro LH, Abdo Bde A, Descio FJ, Martucci CE Jr, Serruya DC. [Nonspecific low back pain in young adults: associated risk factors]. Rev Bras Reumatol. 2014 Sep-Oct;54(5):371-7. doi: 10.1016/j.rbr.2014.03.018. Epub 2014 Jul 6. Portuguese. PMID 25627301
- [Background] Chiarotto A, Maxwell LJ, Ostelo RW, Boers M, Tugwell P, Terwee CB. Measurement Properties of Visual Analogue Scale, Numeric Rating Scale, and Pain Severity Subscale of the Brief Pain Inventory in Patients With Low Back Pain: A Systematic Review. J Pain. 2019 Mar;20(3):245-263. doi: 10.1016/j.jpain.2018.07.009. Epub 2018 Aug 10. PMID 30099210
- [Background] Balague F, Mannion AF, Pellise F, Cedraschi C. Non-specific low back pain. Lancet. 2012 Feb 4;379(9814):482-91. doi: 10.1016/S0140-6736(11)60610-7. Epub 2011 Oct 6. PMID 21982256
- [Background] Seyedhoseinpoor T, Sanjari MA, Taghipour M, Dadgoo M, Mousavi SJ. Spinopelvic malalignment correlates to lumbar instability and lumbar musculature in chronic low back pain-an exploratory study. Sci Rep. 2024 Dec 30;14(1):31974. doi: 10.1038/s41598-024-83570-6. PMID 39738674
- [Background] Celik D, Mutlu EK. Clinical implication of latent myofascial trigger point. Curr Pain Headache Rep. 2013 Aug;17(8):353. doi: 10.1007/s11916-013-0353-8. PMID 23801006
- [Background] Xu A, Huang Q, Rong J, Wu X, Deng M, Ji L. Effectiveness of ischemic compression on myofascial trigger points in relieving neck pain: A systematic review and meta-analysis. J Back Musculoskelet Rehabil. 2023;36(4):783-798. doi: 10.3233/BMR-220045. PMID 36872769
- [Background] Siglan U, Colak S. Effects of diaphragmatic and iliopsoas myofascial release in patients with chronic low back pain: A randomized controlled study. J Bodyw Mov Ther. 2023 Jan;33:120-127. doi: 10.1016/j.jbmt.2022.09.029. Epub 2022 Sep 29. PMID 36775506
- [Background] Desai R, Rathi M, Palekar TJ. Effects of Movement Retraining and Lumbar Stabilization Exercises in Mechanical Low Back Pain: A Pilot Study. Cureus. 2024 Feb 16;16(2):e54291. doi: 10.7759/cureus.54291. eCollection 2024 Feb. PMID 38496129
- [Background] Perret C, Poiraudeau S, Fermanian J, Colau MM, Benhamou MA, Revel M. Validity, reliability, and responsiveness of the fingertip-to-floor test. Arch Phys Med Rehabil. 2001 Nov;82(11):1566-70. doi: 10.1053/apmr.2001.26064. PMID 11689977
- [Background] Liu Y, Palmer JL. Iliacus tender points in young adults: a pilot study. J Am Osteopath Assoc. 2012 May;112(5):285-9. PMID 22582198
- [Background] Takamoto K, Bito I, Urakawa S, Sakai S, Kigawa M, Ono T, Nishijo H. Effects of compression at myofascial trigger points in patients with acute low back pain: A randomized controlled trial. Eur J Pain. 2015 Sep;19(8):1186-96. doi: 10.1002/ejp.694. Epub 2015 Mar 24. PMID 25808188
- [Background] Fernandes WVB, Blanco CR, Politti F, de Cordoba Lanza F, Lucareli PRG, Correa JCF. The effect of a six-week osteopathic visceral manipulation in patients with non-specific chronic low back pain and functional constipation: study protocol for a randomized controlled trial. Trials. 2018 Mar 2;19(1):151. doi: 10.1186/s13063-018-2532-8. PMID 29499728